CLINICAL TRIAL: NCT00311623
Title: A Pharmacodynamic Study of Pre-Prostatectomy Rapamycin in Men With Advanced Localized Prostate Cancer
Brief Title: Sirolimus Before Surgery in Treating Patients With Advanced Localized Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: J0576; P30CA006973 (NIH); CDR0000468942 (Other: other); NA_00001011 (Other: JHM IRB)
Record Dates: First submitted 2006-04-05; First posted 2006-04-06 (Estimated); Results first posted 2019-02-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Prostate Cancer
Keywords: stage III prostate cancer; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Sirolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control group (Active Comparator): Men >18years old with prostate cancer clinical stages T1c to T3, no metastases, Gleason sum of 7-10, multiple positive diagnostic cores, Eastern Cooperative Oncology Group (ECOG) performance status of 0-1, candidates for radical prostatectomy.
  Receive no intervention on Days 1-14. Surgery performed on Day 15.
  Interventions: Procedure: Radical prostatectomy
- Low-dose Rapamycin (3mg) (Experimental): Men >18years old with prostate cancer clinical stages T1c to T3, no metastases, Gleason sum of 7-10, multiple positive diagnostic cores, Eastern Cooperative Oncology Group (ECOG) performance status of 0-1, candidates for radical prostatectomy.
  Must have adequate hepatic, renal and bone marrow function, no allergy to rapamycins, avoid medications interfering with rapamycin metabolism, no active infection, no prior therapies for prostate cancer.
  Will receive rapamycin 3mg (Wyeth Pharmaceuticals, 1mg tablets) oral (PO) once daily on Days 1-14 with the last dose given on the morning before surgery (Day 15).
  Interventions: Drug: Rapamycin 3mg; Procedure: Radical prostatectomy
- High-dose Rapamycin (6mg) (Experimental): Men >18years old with prostate cancer clinical stages T1c to T3, no metastases, Gleason sum of 7-10, multiple positive diagnostic cores, Eastern Cooperative Oncology Group (ECOG) performance status of 0-1, candidates for radical prostatectomy.
  Must have adequate hepatic, renal and bone marrow function, no allergy to rapamycins, avoid medications interfering with rapamycin metabolism, no active infection, no prior therapies for prostate cancer.
  Will receive rapamycin 6mg (Wyeth Pharmaceuticals, 2mg tablets) oral (PO) once daily on Days 1-14 with the last dose given on the morning before surgery (Day 15).
  Interventions: Drug: Rapamycin 6mg; Procedure: Radical prostatectomy

INTERVENTIONS:
Drug: Rapamycin 3mg — Rapamycin 3mg (Wyeth Pharmaceuticals, 1mg tablets) PO once daily on Days 1-14 with the last dose given on the morning before surgery (Day 15).
  Other Names: sirolimus
  Arms: Low-dose Rapamycin (3mg)
Drug: Rapamycin 6mg — Rapamycin 6mg (Wyeth Pharmaceuticals, 2mg tablets) PO once daily on Days 1-14 with the last dose given on the morning before surgery (Day 15).
  Other Names: sirolimus
  Arms: High-dose Rapamycin (6mg)
Procedure: Radical prostatectomy — Radical prostatectomy performed on Day 15

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as sirolimus, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This clinical trial is studying the best dose of sirolimus and to see how well it works before surgery in treating patients with advanced localized prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the pharmacodynamically optimal dose (POD) of continuous daily oral sirolimus (rapamycin) in patients with advanced localized prostate cancer when given prior to radical prostatectomy, as measured by tumor S6 kinase inhibition by immunohistochemistry (IHC).
* Determine the proportion of men with downstream target inhibition in prostate tumor tissue at the POD using paired tumor biopsies from before and after rapamycin administration.
* Correlate tumor pharmacodynamic (PD) efficacy with a surrogate marker of tumor PD efficacy, peripheral blood mononuclear cell (PBMC) S6 kinase activity inhibition.

Secondary

* Characterize the serum and prostate tissue pharmacokinetics of daily oral rapamycin at 2 dose levels.
* Determine the relationship of PD target inhibition of S6 kinase activity with pretreatment Akt activity and PTEN loss by IHC in prostate cancer.
* Describe the relationship between PD inhibition with the mTOR inhibitor rapamycin and pretreatment prostate biopsy Gleason sum, Ki-67 index of proliferation, Akt activity, p27 IHC, and PTEN.
* Correlate PD efficacy as measured by downstream S6 kinase activity inhibition with markers of increased apoptosis (activated caspase 3) and reduction in markers of proliferation (change in Ki-67) in prostate tumor specimens.
* Quantify and characterize the toxicity of daily continuous rapamycin at 2 dose levels in generally healthy men with prostate cancer prior to surgery.
* Evaluate the activity of rapamycin in prostate cancer as measured in prostate specific antigen response prior to surgery.

OUTLINE: This is a multicenter, dose-escalation study.

Patients receive oral sirolimus (rapamycin) once daily on days 1-14 in the absence of unacceptable toxicity.

Cohorts of 12-21 patients receive escalating doses of rapamycin until the pharmacodynamically optimal dose is determined.

Patients undergo radical prostatectomy on day 15.

Patients undergo blood collection and tumor biopsies periodically during study for pharmacologic and correlative biomarker studies.

After completion of study treatment, patients are followed at 30 and 90 days.

PROJECTED ACCRUAL: A total of 42 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically determined adenocarcinoma of the prostate

  * Stage T1c-T3b disease
  * No evidence of disease that has spread beyond the prostate or seminal vesicles
* No metastatic prostate cancer, including bone, visceral, brain, and lymph node metastases
* Tumor Gleason score sum of 7-10 (4+3 and 3+4 allowed) with tumor involving at least 2 discrete core biopsy sections
* Scheduled to undergo radical prostatectomy
* No other subtypes of prostate cancer, including any of the following:

  * Sarcoma
  * Neuroendocrine tumors
  * Small cell cancer
  * Ductal cancer
  * Lymphoma

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* WBC > 3,500/mm^3
* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 100,000/mm^3
* Hemoglobin > 9 g/dL
* Creatinine < 2.0 mg/dL
* Bilirubin < 2 mg/dL
* ALT and AST < 2 times upper limit of normal (ULN)
* Alkaline phosphatase < 2 times ULN
* Triglycerides and total cholesterol < 2 times ULN
* No history of allergy to sirolimus (rapamycin) or its derivatives
* No uncontrolled medical condition that would increase risk or limit compliance with study requirements, including the following:

  * Immunodeficiency
  * Gastrointestinal disease that would limit ability to swallow, take oral medications, or absorb them
* No active infections
* No other concurrent malignancy

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior chemotherapy, biologic therapy, radiotherapy, or immunotherapy for prostate cancer
* No concurrent chronic treatment with immunosuppressants or medications that interfere with the metabolism of sirolimus (rapamycin)
* No concurrent medication or agents that would interfere with the metabolism or excretion of rapamycin or its derivatives, including any of the following:

  * Phenytoin
  * Carbamazepine
  * Cyclosporine
  * Clarithromycin
  * Clotrimazole
  * Erythromycin
  * Amiodarone
  * Protease inhibitors used to treated HIV infection
  * Cisapride
  * Grapefruit juice
  * Diltiazem
  * Tacrolimus
  * Hypericum perforatum (St. John's wort)
  * Barbiturates
  * Rifampin
  * Phenobarbital
  * Rifabutin
  * Efavirenz
  * Nevirapine
* At least 7 days since prior herbal medicines and medications, including any of the following:

  * Hydrastis canadensis (goldenseal)
  * Uncaria tomentosa (cat's claw)
  * Echinacea angustifolia roots
  * Trifolium pretense (wild cherry)
  * Chamomile
  * Glycyrrhiza glabra (licorice)
  * Dillapiol
  * Naringenin
  * Norfloxacin
  * Atorvastatin
  * Pravastatin
  * Cimetidine
  * Fluconazole

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2008-01 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Carducci, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (3):
- United States (3):
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Duke Comprehensive Cancer Center, Durham, North Carolina

REFERENCES:
- [Result] Armstrong AJ, Netto GJ, Rudek MA, Halabi S, Wood DP, Creel PA, Mundy K, Davis SL, Wang T, Albadine R, Schultz L, Partin AW, Jimeno A, Fedor H, Febbo PG, George DJ, Gurganus R, De Marzo AM, Carducci MA. A pharmacodynamic study of rapamycin in men with intermediate- to high-risk localized prostate cancer. Clin Cancer Res. 2010 Jun 1;16(11):3057-66. doi: 10.1158/1078-0432.CCR-10-0124. Epub 2010 May 25. PMID 20501622

RESULTS

PARTICIPANT FLOW:
Groups:
- Control Group: Men >18years old with prostate cancer clinical stages T1c to T3, no metastases, Gleason sum of 7-10, multiple positive diagnostic cores, Eastern Cooperative Oncology Group (ECOG) performance status of 0-1, candidates for radical prostatectomy.
  Receive no intervention on Days 1-14. Surgery performed on Day 15.
  Radical prostatectomy: Radical prostatectomy performed on Day 15
- Low-dose Rapamycin (3mg): Men >18years old with prostate cancer clinical stages T1c to T3, no metastases, Gleason sum of 7-10, multiple positive diagnostic cores, Eastern Cooperative Oncology Group (ECOG) performance status of 0-1, candidates for radical prostatectomy.
  Must have adequate hepatic, renal and bone marrow function, no allergy to rapamycins, avoid medications interfering with rapamycin metabolism, no active infection, no prior therapies for prostate cancer.
  Will receive rapamycin 3mg (Wyeth Pharmaceuticals, 1mg tablets) oral (PO) once daily on Days 1-14 with the last dose given on the morning before surgery (Day 15).
  Rapamycin 3mg: Rapamycin 3mg (Wyeth Pharmaceuticals, 1mg tablets) PO once daily on Days 1-14 with the last dose given on the morning before surgery (Day 15).
  Radical prostatectomy: Radical prostatectomy performed on Day 15
- High-dose Rapamycin (6mg): Men >18years old with prostate cancer clinical stages T1c to T3, no metastases, Gleason sum of 7-10, multiple positive diagnostic cores, Eastern Cooperative Oncology Group (ECOG) performance status of 0-1, candidates for radical prostatectomy.
  Must have adequate hepatic, renal and bone marrow function, no allergy to rapamycins, avoid medications interfering with rapamycin metabolism, no active infection, no prior therapies for prostate cancer.
  Will receive rapamycin 6mg (Wyeth Pharmaceuticals, 2mg tablets) oral (PO) once daily on Days 1-14 with the last dose given on the morning before surgery (Day 15).
  Rapamycin 6mg: Rapamycin 6mg (Wyeth Pharmaceuticals, 2mg tablets) PO once daily on Days 1-14 with the last dose given on the morning before surgery (Day 15).
  Radical prostatectomy: Radical prostatectomy performed on Day 15
Period: Overall Study
Arm/Group | Control Group | Low-dose Rapamycin (3mg) | High-dose Rapamycin (6mg)
Started | 10 | 20 | 2
Completed | 10 | 20 | 0
Not Completed | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Low-dose Rapamycin (3mg) | High-dose Rapamycin (6mg) | Total
Number analyzed (Participants) | 10 | 20 | 2 | 32
Age, Customized [Median (Full Range); unit: years] | 64 [51 to 68] | 61.5 [50 to 81] | 57.5 [51 to 64] | 62.5 [50 to 81]
Sex: Female, Male [Count of Participants; unit: Participants] — All participants were male
  Participants
    Female | 0 | 0 | 0 | 0
    Male | 10 | 20 | 2 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  non-Hispanic | 10 | 20 | 2 | 32
  Caucasian | 10 | 16 | 2 | 28
  African-American | 0 | 4 | 0 | 4
Region of Enrollment [Number; unit: participants]
  United States | 10 | 20 | 2 | 32
Body Mass Index [Median (Standard Deviation); unit: kg/m2] | 28.0 (2.31) | 27.8 (4.95) | 28.7 (1.75) | 27.83 (4.09)
Biopsy Gleason sum [Count of Participants; unit: Participants] — The Gleason sum ranges from 2-10 with a higher score reflecting less-differentiated tumors with worse prognosis. The total is a sum of two numbers which are based on the microscopic appearance of cells. The first number is the score based on the dominant, cell morphology (scored 1-5) and the second number is based on the highest grade of the non-dominant cell pattern (scored 1-5).
  Participants
    6 | 0 | 1 | 0 | 1
    7 | 9 | 17 | 1 | 27
    8-10 | 1 | 2 | 1 | 4
Radical prostatectomy (RP) Gleason sum [Count of Participants; unit: Participants] — The Gleason sum ranges from 2-10 with a higher score reflecting less-differentiated tumors with worse prognosis. The total is a sum of two numbers which are based on the microscopic appearance of cells. The first number is the score based on the dominant, cell morphology (scored 1-5) and the second number is based on the highest grade of the non-dominant cell pattern (scored 1-5).
  Participants
    6 | 3 | 3 | 0 | 6
    7 | 6 | 15 | 2 | 23
    8-10 | 1 | 2 | 0 | 3
Preoperative clinical stage [Count of Participants; unit: Participants] — Clinical stage is estimated based on results of physical exam, biopsy or any imaging tests.
  Staging is defined by the American Joint Committee on Cancer (AJCC) TNM system where T= primary tumor, N= spread to nearby lymph nodes, M= metastasis, Grade Group 1 through 5 (based on Gleason score, higher grade group reflects higher Gleason score), and further letter ("a" through "c" staging. A lower number reflects less spread of cancer and a lower letter reflects a lower stage.
  Participants
    T1c | 6 | 13 | 2 | 21
    T2a | 0 | 4 | 0 | 4
    T2b | 3 | 2 | 0 | 5
    T2c | 1 | 1 | 0 | 2
Pathologic stage [Count of Participants; unit: Participants] — Pathological stage is assessed by analyzing tissue collected from prostatectomy. Staging is defined by the American Joint Committee on Cancer (AJCC) TNM system where T= primary tumor, N= spread to nearby lymph nodes, M= metastasis, Grade Group 1 through 5 (based on Gleason score, higher grade group reflects higher Gleason score), and further letter ("a" through "c" staging. A lower number reflects less spread of cancer and a lower letter reflects a lower stage.
  Participants
    T2 | 6 | 10 | 2 | 18
    T3a | 3 | 7 | 0 | 10
    T3b | 0 | 3 | 0 | 3
    TX N1 | 1 | 0 | 0 | 1
Any PSA Decline [Count of Participants; unit: Participants] — Population: Data for PSA decline was not collected for 5 participants from the Control Arm and 3 participants from the Low-dose arm.
  Participants
    number analyzed (Participants) | 5 | 17 | 2 | 24
    (all) | 1 | 4 | 1 | 6
Preoperative D'Amico risk [Count of Participants; unit: Participants] — Population: Data for Undetectable day 90 PSA was not collected for 5/10 participants from the Control Arm.
  Participants
    Low | 0 | 1 | 0 | 1
    Intermediate | 8 | 17 | 1 | 26
    High | 2 | 2 | 1 | 5
    Undetectable day 90 PSA: number analyzed (Participants) | 5 | 20 | 2 | 27
    Undetectable day 90 PSA | 4 | 17 | 2 | 23

OUTCOME MEASURES:

1. Primary Outcome: Pharmocodynamically Optimal Dose (POD) of Rapamycin as Determined by Number of Participants With Greater Than or Equal to 60% Tumor S6 Kinase Inhibition by Immunohistochemistry (IHC).
Time Frame: Day 15 post-intervention
Population: Only 10 participants from the low-dose arm and 8 participants from the control arm had adequate paired tissue for evaluation, due to the lack of availability or inadequacy of either biopsy or radical prostatectomy. The 2 patients from the high-dose arm did not complete due to dose-limiting toxicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Low-dose Rapamycin (3mg) | High-dose Rapamycin (6mg)
Number analyzed (Participants) | 8 | 10 | 0
Participants | 1 | 5 |

2. Primary Outcome: Median S6 Kinase Inhibition in Prostate Tumor Tissue at the POD
Time Frame: Change from baseline to 15 days post-intervention
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of S6 kinase inhibition
Arm/Group | Control Group | Low-dose Rapamycin (3mg) | High-dose Rapamycin (6mg)
Number analyzed (Participants) | 8 | 10 | 0
percentage of S6 kinase inhibition | 2 [-6 to 30] | 58 [-15 to 82] |

3. Primary Outcome: Pharmacodynamic Response as Assessed by Median Post-treatment S6 Activity H-score
Description: Pharmocodynamic response was taken as ≥60% decrease in the H-score for S6 phosphorylation in the radical prostatectomy tumor tissue compared with the pretreatment (baseline) biopsy tumor tissue. The H-score is a semiquantitative measure of the percentage of cells scoring positive (0-100) multiplied by the intensity of staining (0-3).
Time Frame: Change from baseline to 15 days post-intervention
Population: Only 9 participants from the control group and 13 participants in the low-dose arm had evaluable tissue for analysis. Participants in the high dose arm did not complete the study due to serious adverse events.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Control Group | Low-dose Rapamycin (3mg) | High-dose Rapamycin (6mg)
Number analyzed (Participants) | 9 | 13 | 0
score on a scale | 140 [NA to NA] — Original data to report a dispersion measure cannot be located. | 70 [NA to NA] — Original data to report a dispersion measure cannot be located. |

4. Secondary Outcome: Pharmacokinetic Response of Rapamycin 3mg as Assessed by Whole Blood Analysis
Description: Snap-frozen prostate tissue was evaluated for tissue rapamycin levels.
Time Frame: Change from baseline to 15 days post-intervention
Population: Data was not collected for this outcome measure
Arm/Group | High-dose Rapamycin (6mg)
Number analyzed (Participants) | 0

5. Secondary Outcome: Pharmacokinetic Response of Rapamycin 6mg as Assessed by Whole Blood Analysis
Description: Snap-frozen prostate tissue was evaluated for tissue rapamycin levels.
Time Frame: Change from baseline to 15 days post-intervention
Population: 0/2 participants tolerated this dose. Therefore, data for this outcome measure was not collected.
Arm/Group | High-dose Rapamycin (6mg)
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants With Change in Akt Phosphorylation as Measured by Immunohistochemistry (IHC)
Description: Number of participants with change (increased, decreased or no change) in Akt phosphorylation as measured by immunohistochemistry (IHC)
Time Frame: Change from baseline to 15 days post-intervention
Population: Only 7 participants from the control group and 10 participants in the low-dose arm had adequate paired tissue for analysis. Participants in the high dose arm did not complete the study due to serious adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Low-dose Rapamycin (3mg) | High-dose Rapamycin (6mg)
Number analyzed (Participants) | 7 | 10 | 0
Participants
  increased AKT phosphorylation | 3 | 4 |
  decreased AKT phosphorylation | 3 | 4 |
  no change in AKT phosphorylation | 1 | 2 |

7. Secondary Outcome: PTEN Loss as Measured by Immunohistochemistry (IHC)
Description: Determine the relationship of PD target inhibition of S6 kinase activity with pretreatment PTEN loss by IHC in prostate cancer.
Time Frame: Change from baseline to 15 days post-intervention
Population: Data was not collected for this outcome measure
Arm/Group | Control Group | Low-dose Rapamycin (3mg) | High-dose Rapamycin (6mg)
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: p27 as Measured by Immunohistochemistry (IHC)
Description: p27 by IHC in prostate cancer.
Time Frame: Change from baseline to 15 days post-intervention
Population: Data was not collected for this outcome measure
Arm/Group | Control Group | Low-dose Rapamycin (3mg) | High-dose Rapamycin (6mg)
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Change in Gleason Sum
Description: pretreatment biopsy compared to post-treatment radical prostatectomy specimen
Time Frame: Change from baseline to 15 days post-intervention
Population: Data was not collected for this outcome measure
Arm/Group | Control Group | Low-dose Rapamycin (3mg) | High-dose Rapamycin (6mg)
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Increased Apoptosis as Measured by Activated Caspase 3
Description: Correlate PD efficacy as measured by downstream S6 kinase activity inhibition with markers of increased apoptosis (activated caspase 3) in prostate tumor specimens.
Time Frame: Baseline, 14 days post-intervention, 90-days post-operative
Population: Data was not collected for this outcome measure
Arm/Group | Control Group | Low-dose Rapamycin (3mg) | High-dose Rapamycin (6mg)
Number analyzed (Participants) | 0 | 0 | 0

11. Secondary Outcome: Reduction in Proliferation as Measured by Decrease in Ki-67
Description: Correlate PD efficacy as measured by downstream S6 kinase activity inhibition with markers of reduction in markers of proliferation (change in Ki-67) in prostate tumor specimens.
Time Frame: Baseline, 14 days post-intervention, 90-days post-operative
Population: Data was not collected for this outcome measure
Arm/Group | Control Group | Low-dose Rapamycin (3mg) | High-dose Rapamycin (6mg)
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Toxicity as Per National Cancer Institute Common Toxicity Criteria v3.0
Description: Dose-limiting toxicity was defined as grade 3/4 neutropenia with fever lasting >7 days, platelets of <100,000/mm3 or associated with bleeding, grade ≥3 non-hematologic toxicity, or irreversible grade 2 toxicity related to rapamycine.
Time Frame: Baseline, 14 days post-intervention, 90-days post-operative
Population: Data was not collected for this outcome measure
Arm/Group | Control Group | Low-dose Rapamycin (3mg) | High-dose Rapamycin (6mg)
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Activity of Rapamycin as Measured by Prostate Specific Antigen (PSA) Response Prior to Surgery
Description: PSA response to daily rapamycin
Time Frame: Change from baseline to Day 14
Population: Data was not collected for this outcome measure
Arm/Group | Control Group | Low-dose Rapamycin (3mg) | High-dose Rapamycin (6mg)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Day 90 post-operative
Arm/Group | Control Group | Low-dose Rapamycin (3mg) | High-dose Rapamycin (6mg)
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/20 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/20 | 2/2
Other Adverse Events (participants affected / at risk) | 1/10 | 8/20 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Group (N=10) | Low-dose Rapamycin (3mg) (N=20) | High-dose Rapamycin (6mg) (N=2)
Severe thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Control Group (N=10) | Low-dose Rapamycin (3mg) (N=20) | High-dose Rapamycin (6mg) (N=2)
Post-operative ileus (Surgical and medical procedures) | 1 | 2 | 0
Maculopapular rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 0 — Grade 1-2 Neutropenia without fever
Stomatitis (Infections and infestations) | 0 | 2 | 2
Fever (Immune system disorders) | 0 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 — Grade 1 thrombocytopenia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes